CLINICAL TRIAL: NCT04886336
Title: The Impact of Tenofovir Alafenamide on Profiles of Body Weight and Metabolic Features in Chronic Hepatitis B Patients
Acronym: HBV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-ER 109-100
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2020-07

CONDITIONS: HBV
Keywords: Body Weight; Metabolic; Tenofovir alafenamide
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Biospecimen Retention: Samples Without DNA — We collection plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tenofovir Disoproxil Fumarate(TDF) switch to TAF: The indications of TDF switching to TAF due to adverse events of TDF or physician's judgement according to clinical conditions.
- Entecavir(ETV)switch to Tenofovir Alafenamide(TAF): In entecavir switch group, at least 30 patients should have baseline BW data before entecavir treatment. The indications of entecavir switching to TAF include suboptimal HBV suppression (defined as detectable HBV DNA after at least one year of entecavir treatment), adverse events due to entecavir, physician's judgement according to clinical conditions.
- observation groups with take either entecavir (25patients) or TDF (25 patients).: observation groups with total 50 patients who continuously take either entecavir (25patients) or TDF (25 patients) will be enrolled.Examination schedules for these two additional groups are the same as switching groups.

SUMMARY:
The aim of this study is to compare the BW and metabolic profiles of CHB patient before and after shifting to TAF therapy.

In this study, investigators will enroll 100 entecavir and 100 TDF treated CHB patients who will switch to TAF and then follow for one year. Demographic, liver function tests, sugar profiles, lipid profiles, ASCVD risk score, body weight, body weight, body height, and waist circumference will be checked and recorded periodically.

Investigators anticipated that body weight will change significantly after switching to TAF in both entecavir and TDF group and may associated with increased risk of cardiovascular risk.

DETAILED DESCRIPTION:
Currently, three oral nucleoside/tides analogues (NUC), including entecavir(ETV), tenofovir disoproxil fumarate (TDF), and tenofovir alafenamide (TAF), are available as the first line of treatment option for chronic hepatitis B (CHB) in Taiwan. Among them, TDF exhibits a greater decline of cholesterol, High-density lipoprotein(HDL), and low-density lipoprotein (LDL) levels than entecavir, while the impact of such general lipid-lowering effects on the risk of atherosclerotic cardiovascular diseases (ASCVD) remains unclear. For metabolic features, the evidence comes from HIV patients treated with TDF or TAF containing anti-retroviral therapy (ART). In one study revealed that a 0.45 kg/m2 increase of body mass index (BMI) and a 13% of increase in ASCVD risk score after switching from TDF-containing to TAF-containing ART. Weight gain after starting ART has been reported to associate with lower mortality in initial under-weight or normal-weight HIV patients. However, a study compared the efficacy and safety of dolutegravir/TAF/emtricitabine, dolutegravir/TDF/emtricitabine, and EFV/TDF/emtricitabine and revealed that patients receiving TAF and TDF containing regimens significantly increased body weight. The subsequent body composition analysis showed weight gain mainly resulted from increased lean muscle and fat of trunk and limb. A previous study also showed that the ART-associated increase in muscle area, regardless of regimen, is likely a reflection of increased fat within the muscle that may associate with weakness of muscle strength, risk of fall, and a decline of physical activities.

Overall, in HIV-infected patients, TAF-containing regimens had been shown to increase body weight resulting from increased fat and muscle of trunk and limb. However, it remains unknown whether all these findings in HIV infected patients could be similarly observed in CHB patient receiving TAF therapy, which is commonly encountered in Asia-Pacific region. Moreover, the mechanisms underlying these changes are still unclear. The long-term clinical impact of the BW gain and associated metabolic derangement is also unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 20 years.
2. Chronic hepatitis B virus infection defined as presence of positive HBsAg more than 6 months.
3. TAF naïve.
4. Patients already receiving TDF or entecavir treatment, and the scheduled NUC treatment from enrolment being greater than one year.

Exclusion Criteria:

1. Other etiology of chronic hepatitis.
2. Severe comorbid disorders.
3. Patients with History of acute coronary syndrome, myocardial infarction, stable angina, coronary/other arterial revascularization, stroke, transient ischemic attack, or peripheral arterial disease from atherosclerosis.
4. Uncontrolled diabetes mellitus (HBA1c > 8.5%).
5. Current evidence or suspicious of malignancy.
6. eGFR <50 ml/min/1.73m2.
7. Any one of following hematology or biochemical or clinical abnormalities indicating the presence of liver decompensation: Albumin <3.5g/dL, Total Bilirubin >2.5mg/dL, prothrombin time prolongation >4 sec or INR >1.7, platelet count <100 x 103 uL, and history or presence of ascites or hepatic encephalopathy.
8. Child-bearing age women without the willing to contraceptive control, or lactating or pregnant women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients who have been treated with TDF (n=100) or entecavir (n=100) will switch to TAF.
  In entecavir switch group, at least 30 patients should have baseline BW data before entecavir treatment. The indications of entecavir switching to TAF include suboptimal HBV suppression (defined as detectable HBV DNA after at least one year of entecavir treatment), adverse events due to entecavir, patient's decision, and physician's judgement according to clinical conditions.
  The scheduled treatment duration from enrolment should be greater than one year. Treatment indications for HBeAg-positive chronic hepatitis B, HBeAg-negative chronic hepatitis B and liver cirrhosis are based on reimbursement criteria of Taiwan government.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
1.Body weight changes after shifting to TAF treatment. | 48 weeks
  Collection Body weight data before and after treatment.

SECONDARY OUTCOMES:
2.Changes of lipid and sugar profiles before and after shifting to TAF treatment. | 48 weeks.
  Collection lipid( include TG<mg/dl>/Chol<mg/dl>,/LDL<mg/dl>/ HDL<mg/dl>) data and sugar profiles(include Insulin<uU/ml>, fasting sugar<mg/dl>, glycosylated hemoglobin<%>) data before and after treatment.
3.Virologic responses following TAF treatment. | 48 weeks.
  Collection Virologic data (e.g HBV DNA<IU/ml>,)before and after treatment.
4.Renal function after shifting to TAF treatment. | 48 weeks.
  Collection Renal function(include Cr<mg/dL>/eGFR<ml/min/1.73m2>)data before and after treatment.
5. ASCVD score changes before and after shifting to TAF treatment. | 48 weeks.
  Collection ASCVD score before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Nan Cheng, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan